CLINICAL TRIAL: NCT02214030
Title: A Randomized Comparison of Assiut Femoral Compression Device Versus Manual Compression in the Achievement of Hemostasis After Percutaneous Coronary Intervention
Brief Title: Efficacy Study of Assiut Femoral Compression Device Versus Manual Compression in the Achievement of Hemostasis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman khairy Mohamed, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFCD-03; AUH-03 (Other: Assiut University)
Record Dates: First submitted 2014-07-26; First posted 2014-08-12 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Common Femoral Artery Injury; Other Vascular Adverse Event
Keywords: Femoral compression device; manual compression; arterial hemostasis; coronary intervention; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assiut Femoral Compression Device (Active Comparator): the sheaths were removed 2 hours after PCI instead of conventional 6hours. To standardize compression times, AFCD were applied to patient and complete femoral artery compression were applied for 5 minutes, followed by a gradual release of pressure over the ensuing 8 minutes. Therefore each patient received a minimum of 13 minutes of compression, with further compression applied only if full hemostasis had not been achieved at that point with maximum of 30 minutes.
  Interventions: Device: Assiut Femoral Compression Device
- Manual compression (Placebo Comparator): The intra-arterial sheaths were removed 6 hours after PCI in the MC group according to the standard local protocols.
  Interventions: Device: Assiut Femoral Compression Device

INTERVENTIONS:
Device: Assiut Femoral Compression Device — Assiut Femoral Compression Devices (AFCD) is a femoral compression system, The pressure dome is situated over the vessel puncture site in the groin and applies a mechanical pressure over the vessel puncture site to induce hemostasis.
  Other Names: AFCD

SUMMARY:
This study was performed to evaluate the safety and efficacy of a locally designed Assiut Femoral Compression Device (AFCD) versus manual compression (MC). Femoral compression devices have been developed thorough the past decades without being strongly implemented in the catheterization laboratory. Their limited adoption reflects concerns of high cost and conflicting data regarding their safety

DETAILED DESCRIPTION:
The intra-arterial sheaths were removed 6 hours after PCI in the MC group according to the standard local protocols. However for AFCD group, the sheaths were removed 2 hours after PCI instead of conventional 6 hours. To standardize compression times, AFCD were applied to patient and complete femoral artery compression were applied for 5 minutes, followed by a gradual release of pressure till distal pulse is palpated. Each patient received a minimum of 13 minutes of compression, with further compression applied only if full hemostasis had not been achieved at that point with maximum of 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 85 years of age,
* Scheduled to undergo an elective PCI via arterial puncture of common femoral artery were eligible for enrollment in the study.
* Elective PCI was defined as any coronary revascularization in a low-risk patient who presents to the facility for a planned PCI or for a coronary angiogram followed by ad hoc PCI.

Exclusion Criteria:

Patients were excluded from the study if the patient has

1. Any procedural complication included:

   * prolonged chest pain,
   * transient coronary artery closure, no-flow or slow-flow phenomenon,
   * hemodynamic instability,
   * persistent electrocardiographic changes,
   * side-branch occlusion of >1.5 mm, or
   * an angiographically suboptimal result,
2. Arterial access other than the right or left femoral artery ,
3. Vascular perforation, thrombosis during procedure ,
4. Patients with high risk of puncture site complications as:

   * Bleeding diathesis,
   * International normalized ratio >1.5,
   * Recent thrombolysis,
   * Low platelet count,
   * Hematoma at the end of the procedure,
   * Previous iliofemoral artery surgery or any peripheral vascular Surgery,
   * Previous femoral artery complication from angiography, and
5. Uncontrolled hypertension at time of procedure (>180/>110).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time-To-Ambulation (TTA), measured in hours | TTA was measured from the time the introducer sheath was removed (2 hr in AFCD group and 6 hours in MC group after end of PCI) to time of ambulation
  Ambulation was defined as patient standing and walking at least 6 meters (20 feet) without re-bleeding or significant oozing requiring manual compression
the absence of major adverse events on discharge | 24 post procedure
  major adverse event (MAE) was defined as symptomatic bleeding associated with hemoglobin drop ≥5 g/dL requiring blood transfusion, fatal bleeding that directly results in death, a pseudoaneurysm or arteriovenous fistula, distal arterial embolism, infections requiring administration of IV antibiotics or debridement, and the need for vascular surgery.

SECONDARY OUTCOMES:
Device success: | 5 minutes during application
  This was defined as easy application of the device with good fixation and stability and achieving final hemostasis. Device Stability was defined as absence of tilt and/or mobility after application of the device on top of the patient groin. Assessment of the device application was performed using a questionnaire with a scale of three grades; "Easy", "Difficult" and "Requires Improvement". Assessment of stability and fixation of the device was performed on a scale defined as "Very Good", "Good" and "Bad".
Procedure success | 24 h post procedure
  This was defined as hemostasis achieved by the assigned method, without the occurrence of a closure-related major adverse event (MAE).

OTHER OUTCOMES:
Time-To-Hemostasis (TTH), measured in minutes. | TTH was measured from the time the introducer sheath was removed (2 hr in AFCD group and 6 hours in MC group after end of PCI) to the time hemostasis was achieved
  Hemostasis was defined as no or minimal subcutaneous oozing and the absence of expanding or developing hematoma
Minor complications: | 24h post procedure
  Any oozing (leakage of blood from the puncture site requiring digital pressure), ecchymosis (bleeding into subcutaneous tissue planes causing bluish-purple discoloration > 4cm in diameter), hematoma (non pulsatile mass > 1 cm in diameter), and infections treatable with oral antibiotics
Patient discomfort: | within 10 minutes of device application
  was assessed based on a short form of the McGill Pain Questionnaire using a Present Pain Intensity (PPI) scale that rated pain from 0 (no pain) to 5 (excruciating).
Vasovagal manifestations | within 10 minutes of device application
  (sweating, bradycardia, nausea and vomiting) were recorded.
Time the patient is deemed eligible for hospital discharge | within 24 hours post procedure
  Time the patient is deemed eligible for hospital discharge based on the report of the attending resident

CONTACTS AND LOCATIONS:
Overall Officials: Ayman K.M. Hassan, MD. PhD., Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Hassan AKM, Hasan-Ali H, Ali AS. A new femoral compression device compared with manual compression for bleeding control after coronary diagnostic catheterizations. The Egyptian Heart Journal. 2013 (in-press).